CLINICAL TRIAL: NCT07368946
Title: A Pilot Feeding Study to Assess Phosphate Overload in Patients With Chronic Kidney Disease
Brief Title: Phosphate Assessment in Chronic Kidney Disease Patients Study
Acronym: PACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jing Chen, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2024-1240; 68418 (Other: UT Southwestern Medical Center)
Record Dates: First submitted 2025-11-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (Stage 3-4); Chronic Kidney Disease Mineral and Bone Disorder
Keywords: chronic kidney disease; study diet; feeding study; pilot; oral phosphate feeding
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Kidney Disease Patients (Active Comparator): Participants with eGFR >15 ml/min/1.73m2 - < 60 ml/min/1.73m2 for the CKD group
  Interventions: Dietary Supplement: Dietary Phosphorus Intake
- Control Group (Active Comparator): Healthy participants without CKD eGFR ≥ 60 ml/min/1.73m2
  Interventions: Dietary Supplement: Dietary Phosphorus Intake

INTERVENTIONS:
Dietary Supplement: Dietary Phosphorus Intake — Dietary phosphorus intake of about 777 mg/day for 7 days, followed by an increase to about 1,277mg/day for another 7 days, and a further increase to about 1,777 mg/day for the subsequent 7 days.
  The meal plan will maintain consistent intake of calories, sodium, potassium, and calcium throughout the 21-day intervention.
  1200 mg/day and 1700 mg/day phosphorus diets will be achieved by providing participants with sodium phosphate capsules and 777 mg/day meals.

SUMMARY:
The proposed pilot feeding study aims to explore novel pathways in phosphate metabolism and identify new biomarkers, as well as to develop a compound index for assessing phosphate overload with high validity and reliability.

Investigators will address the following specific aims: 1). To explore novel pathways of phosphate metabolism and assess the influence of CKD status on these metabolic pathways. 2). To identify novel biomarkers for phosphate overload that reflect changes in dietary phosphorus intake. 3). To develop a compound phosphate overload index that measures dietary phosphorus intake with high validity and reliability.

This study will provide novel insights into phosphate metabolism and the assessment of phosphate overload in CKD patients. This investigation aims to provide preliminary data to further studies for the development of reliable biomarkers in CKD patients, which could contribute significantly to early interventions and improve health outcomes.

DETAILED DESCRIPTION:
Specifically, study team propose recruiting 30 participants with CKD and 30 without CKD to investigate the responses of blood metabolites and known biomarkers to a 21-day diet intervention. The intervention will consist of a dietary phosphorus intake of about 777 mg/day for 7 days, followed by an increase to about 1,277mg/day for another 7 days, and a further increase to about 1,777 mg/day for the subsequent 7 days. 1200 mg/day and 1700 mg/day phosphorus diets will be achieved by providing participants with sodium phosphate capsules and 777 mg/day meals. The meal plan will maintain consistent intake of calories, sodium, potassium, and calcium throughout the 21-day intervention. Sodium, calcium, and potassium content will not change significantly throughout the intervention. The overnight fasting blood and 24-hour and random urine samples will be collected at the baseline and end of each phase.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years or older, of any race/ethnicity
* Women must either be post-menopausal or have no monthly menstrual cycle
* Estimated total daily energy expenditure (TDEE) of 1700 - 2700 calories
* eGFR >15 ml/min/1.73m2 - < 60 ml/min/1.73m2 for the CKD group (CKD Stage 3 or Stage 4)
* eGFR ≥ 60 ml/min/1.73m2 and negative urine protein on dipstick test for the non-CKD group
* English speaking

Exclusion Criteria:

* Pregnant, currently breastfeeding, or <3 months postpartum
* Current dialysis or kidney transplant patient
* Current use of insulin or chemotherapy drugs
* Smokes cigarettes or uses e-cigarettes (vapes)
* Uses nicotine products or other recreational drugs
* Medical history of stroke or myocardial infarction (MI)
* Medical history of conditions that can affect phosphate metabolism (i.e., uncontrolled thyroid disorder, parathyroid disorder, or gastrointestinal malabsorption disorders [Crohn's, ulcerative colitis, and celiac disease], cirrhosis)
* Current use of certain medications that directly alter phosphate levels (i.e., phosphate binders; phosphate supplements, irregular use of iron)
* Regular use of laxatives
* Hypo- or hyperphosphatemia (serum phosphate < 2.5 or > 4.6 mg/dl)
* Hypo- or hypercalcemia (serum calcium < 8.4 or > 10.7 mg/dl)
* Severe anemia (hemoglobin < 8 g/dl for women and < 9 g/dl for men)
* Severe hyperglycemia (serum blood glucose > 300 mg/dl)
* Body weight less than <110 lbs (due to risk for phlebotomy-induced anemia)
* Received a blood transfusion in the last four months
* Extreme hypertension as demonstrated by a blood pressure > 180/120 as the average of 3 blood pressures taken during the screening/baseline, or extremely low blood pressure < 80/50
* Unwilling or unable to eat study meals
* Lack of access to a functional refrigerator or freezer
* Lack of access to a microwave or conventional oven
* On low potassium diet
* On low phosphate diet
* Specific dietary restrictions (i.e. vegetarian, vegan, ketogenic, etc.)
* Food allergies including but not limited to milk, egg, soy, nuts, shellfish, and wheat or gluten
* Allergic to sodium phosphate
* Unable or unwilling to complete urinary sample collection or food diaries
* Unable or unwilling to provide informed consent
* Unable to read or speak English
* Participant in other conflict clinical trial
* Unable to complete the study measurements
* Unsafe to participate in this study per investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum phosphate levels | Baseline, week 1, week 2, and week 3
  Circulating serum phosphate levels (mg/dL) will be measured using standard clinical laboratory assays
Change in parathyroid hormone (PTH) levels | Baseline, week 1, week 2, and week 3
  Circulating PTH levels (pg/mL) will be measured using standard clinical laboratory assays
Change in C-terminal Fibroblast Growth Factor 23 (FGF23) levels | Baseline, week 1, week 2, and week 3
  Circulating C-terminal FGF23 levels (RU/mL) will be measured using standard clinical laboratory assays
Change in Fibroblast Growth Factor 23 (FGF23) levels | Baseline, week 1, week 2, and week 3
  Circulating FGF23 levels (pg/mL) will be measured using standard clinical laboratory assays
Phosphate burden indices | Baseline, week 1, week 2, week 3
  Phosphate burden indices, developed using machine learning methods to systematically incorporate both known biomarkers and novel biomarkers. No units have been identified, we anticipate creating a score.

SECONDARY OUTCOMES:
Change in serum calcium levels | Baseline, week 1, week 2, and week 3
  Circulating serum calcium levels (mg/dL) will be measured using standard clinical laboratory assays
Change in Alkaline Phosphatase (ALP) levels | Baseline, week 1, week 2, and week 3
  Circulating serum ALP levels (U/L) will be measured using standard clinical laboratory assays
Change in 1,25-dihydroxyvitamin D levels | Baseline, week 1, week 2, and week 3
  Circulating serum 1,25-dihydroxyvitamin D levels (pg/mL) will be measured using standard clinical laboratory assays
Change in Bone-Specific Alkaline Phosphatase (BALP) levels | Baseline, week 1, week 2, and week 3
  Circulating serum BALP levels (U/L) will be measured using standard clinical laboratory assays
Change in urinary calcium levels | Baseline, week 1, week 2, and week 3
  Circulating urinary calcium excretion levels (mg/day) will be measured using standardized laboratory urine assays
Change in urinary phosphorus levels | Baseline, week 1, week 2, and week 3
  Circulating urinary phosphorus excretion levels (mg/day) will be measured using standardized laboratory urine assays

OTHER OUTCOMES:
Exploratory: Phosphate-related biomarkers identified using proteomics platforms | Baseline, week 1, week 2, week 3
  For the proteomics analysis, only novel biomarkers associated with the phosphate diet will be reported, and their quantitative values are expressed as relative fluorescence units (RFU).
Exploratory: Phosphate-related biomarkers identified using metabolomics platforms | Baseline, week 1, week 2, week 3
  For the metabolomic analysis, only novel biomarkers associated with the phosphate diet will be reported. These features are not yet chemically identified, quantitative results are expressed as relative abundances.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IRB approval is required before sharing IPD.
Supporting Information: Study Protocol